CLINICAL TRIAL: NCT07026877
Title: A Prospective, Multicenter, Non-Blinded, Non-Randomized Pivotal Study of the Fenestrated TREO Stent-Graft System in Subjects With Abdominal Aortic Aneurysms Requiring a Fenestrated Graft and Suitable for Endovascular Repair
Brief Title: Endovascular Repair With Fenestrated TREO Stent-Graft System in AAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-0022-24
Record Dates: First submitted 2025-05-28; First posted 2025-06-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Abdominal Aortic Aneurysms (AAA)
Keywords: Abdominal Aortic Aneurysm; juxtarenal; endovascular
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Stage 1 - Roll-in Arm (Experimental): Minimum of 20 subjects (up to 30) with juxtarenal Abdominal Aortic Aneurysm (AAA), being treated with the Fenestrated TREO Stent-Graft System
  Interventions: Device: Fenestrated TREO Stent Graft System

INTERVENTIONS:
Device: Fenestrated TREO Stent Graft System — The Fenestrated TREO Stent-Graft System is a modular, endoluminal, over-the-wire system intended for the endovascular treatment of juxtarenal and pararenal to paravisceral aneurysms requiring a fenestrated stent-graft and having suitable morphology. The system is composed of the following components:
  Fenestrated TREO Bifurcate Stent-Graft - The main body fenestrated bifurcate provides the following; proximal seal, fenestrations and gates for connection to the leg extensions.
  Bridging Stents - The bridging stent connects the main body bifurcated device to the target visceral artery allowing the target anatomy to maintain perfusion while keeping the pathology sealed
  TREO Leg and Straight Extension Stent-Grafts: The Leg Extension and Straight Extension stent-grafts are used to complete coverage of the pathology from the main body bifurcated device to the distal landing zones (usually the common iliac artery just proximal to the iliac bifurcation).

SUMMARY:
The goal of this clinical trial is to learn if the Fenestrated TREO Stent-Graft System works to treat abdominal aneurysms in adults. An abdominal aneurysm is a bulge in the main blood vessel (the aorta) which carries blood from the heart, through the chest and abdomen. It will also learn about the safety of Fenestrated TREO Stent-Graft System.

The main question it aims to answer is: Can the the Fenestrated TREO Stent-Graft System be used to treat participants with a specific type of abdominal aneurysm called a juxtarenal abdominal aortic aneurysm?

Participants will: Have the the Fenestrated TREO Stent-Graft System implanted via an endovascular surgical procedure and visit the hospital for a follow up period of 5 years, for checkups, tests and imaging scans.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of consent
* Life expectancy is greater than 2 years
* An abdominal aortic or aorto-iliac aneurysm requiring a fenestrated graft and with morphology suitable for endovascular repair (confirmed by Computed Tomography (CT) with contrast performed within 6 months of planned implant procedure) as follows:

  1. Maximum aneurysm diameter of ≥5.5 cm for male ( ≥5.0 cm for female) or
  2. Maximum AAA diameter exceeding two times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements (or saccular aneurysm that warrants treatment in the opinion of the investigator) or
  3. Aneurysm with a history of growth > 0.5 cm in 6 months and
  4. Minimum 0 mm of healthy aorta* below the most inferior renal artery that the physician plans on preserving and no renal artery involvement (juxtarenal aneurysms) or
  5. At least one renal artery involved in the aneurysm and minimum 2 mm below the celiac (suprarenal aneurysms) *Healthy aorta is defined as segment of aorta with parallel aortic wall with minimal (<10%) or no difference in diameter and minimal atherosclerotic debris, thrombus, or calcification.
* Proximal landing zone:

  1. ≥20 mm length
  2. 20-32 mm diameter
  3. ≤60° angle relative to the axis of the suprarenal aorta
  4. ≤60° angle relative to the long axis of the aneurysm
* Distal (iliac) landing zone with:

  1. 8-13 mm inside diameter/ ≥10 mm length
  2. >13-20 mm inside diameter/ ≥15 mm length
* Distal aortic diameter (above the iliac bifurcation) ≥70% of the sum of the iliac limb graft diameters
* Minimum 20 mm aortic lumen diameter at the level of the fenestrations
* Pathology that requires maximum 5 fenestrations in the main body
* Pathology that requires fenestration a minimum 3 mm apart (edge to edge)
* Branch vessels (to be bridged to the fenestrated graft) with:

  1. 5-9 mm diameters
  2. ≥13 mm distal landing zone (or ≥15 mm if there is a gap between fenestration and target vessel)
* Adequate renal function to tolerate contrast-enhanced CTA
* Adequate vascular access compatible with required delivery systems
* Willingness to comply with the follow-up evaluation schedule documented in a signed informed consent prior to implant

Exclusion Criteria:

* Pregnant or lactating
* Dissection in abdominal aorta, ruptured aneurysm, or symptomatic aneurysm (as determined by treating physician)
* Implant procedure as planned does not allow for at least one patent hypogastric artery left intact, unless both are occluded on pre-op imaging.
* A branch vessel(s) that is dissected or has significant calcification, tortuosity, thrombus formation that would interfere with bridging stent delivery or sealing (as determined by treating physician)
* Severe untreated coronary artery disease and/or unstable angina, significant areas of myocardium at risk (based on coronary angiogram or radionuclide scans), left ventricular ejection fraction <20%, or recent diagnosis of congestive heart failure (CHF; as determined by treating physician).
* Stroke or myocardial infarction within 6 months of the planned treatment date
* Chronic obstructive pulmonary disease requiring routine need for oxygen therapy outside the hospital setting (e.g., daily or nightly home use)
* Chronic Kidney Disease (CKD) stage ≥3b.*

  * During Stage 2, patients with severe CKD (stage ≥3b) can be included in the Expanded Access Arm if otherwise eligible.
* Active systemic infection or is suspected of having an active systemic infection (e.g., acquired immune deficiency syndrome (AIDS)/human immunodeficiency virus (HIV), sepsis)
* Clinical conditions that would severely compromise or impair x-ray visualization of the aorta (as determined by treating physician).
* History of an aortopathic connective tissue disease (e.g., Marfan's syndrome)
* Mycotic aneurysm
* Significant or circumferential calcification or mural thrombus (as determined by treating physician):

  1. in the proximal aortic neck
  2. in the distal iliac landing zone
  3. within the treatment length, which may adversely impact device patency
* Cannot receive intraprocedural anticoagulation per the investigator's standard of care, or antiplatelet therapy post-procedurally as per the investigator's standard of care.
* Blood coagulation disorder or bleeding diathesis, the treatment for which cannot be suspended pre- and post-repair
* An investigational study drug or biologic within 30 days of planned procedure or an investigational device within one year of planned procedure or any other treatment that may interfere with the interpretation of the study results.
* Medical, social or psychological issues that the investigator believes may interfere with study treatment or follow-up.
* Untreatable allergy or sensitivity to contrast media, nitinol/nickel, Tantalum, Platinum Iridium (PtIr), 316 stainless steel, ePTFE (expanded polytetrafluoroethylene), PTFE (polytetrafluoroethylene) Impregnated polyester fiber, or polyester
* Other major surgical or medical intervention within 45 days of the planned procedure or plan to undergo other major surgical or medical intervention within 45 days post implantation (e.g., coronary artery bypass graft (CABG), organ transplantation, renal stenting)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-05-29 (Estimated); Study Completion 2030-05-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with absence of a major adverse event (Primary Safety Endpoint) | 30-day post-procedure
  The primary safety endpoint is the absence of a major adverse event (MAE) at 30-day post procedure.
  MAEs are defined as follows:
  * All-cause mortality, defined as death due to any cause
  * Myocardial infarction (new onset) based on the Society for Cardiovascular Angiography & Interventions (SCAI) definition
  * Respiratory failure requiring prolonged (>24 hours from anticipated) mechanical ventilation or reintubation
  * Renal function decline resulting in >50% reduction from baseline estimated glomerular filtration rate (eGFR) or new-onset dialysis
  * Bowel ischemia requiring surgical resection or not resolving with medical therapy
  * Disabling stroke (modified Rankin Scale (mRS) score ≥2 at 90 days post event and an increase in ≥1 mRS category from an individual's pre-stroke baseline, as direct result of the neurological event)
  * Paraplegia (grade 3, Society for Vascular Surgery (SVS) Thoracic Endovascular Aortic Repair (TEVAR) guidelines)
Proportion of patients with successful aneurysm treatment through 12-months post-implant procedure (Primary Effectiveness Endpoint) | 12 months post-procedure
  The primary effectiveness endpoint is the proportion of patients with successful aneurysm treatment through 12-months post-implant procedure, which is a composite of technical success and absence of the following:
  * Aneurysm-related mortality: Death occurs within the first 30-days of the index procedure or a secondary intervention, OR any death that results from aneurysm rupture or an aorta-related complication (e.g., implant infection, occlusion, dissection)
  * Aneurysm rupture: Rupture of the native aneurysm sac (treated lesion)
  * Type I/III Endoleak
  * Aneurysm Expansion (>5 mm)
  * Migration (>10 mm)
  * Loss of patency (i.e., complete occlusion of the aortic implant and/or bridging stent(s))
  * Conversion to open surgical repair: Explant of the investigational device due to any cause
  * Secondary intervention (clinically significant) to address loss of patency, fixation or seal
Successful delivery and deployment of the aortic stent-graft and all modular stent-graft components (Technical Success) | Evaluated 30-days post procedure
  Composite:
  * Successful access to the arterial system using remote arterial exposure, percutaneous technique, or open surgical conduit without the need for unanticipated corrective intervention related to access
  * Successful delivery and deployment of the aortic stent-graft and all modular stent-graft components without the need for unanticipated corrective intervention related to delivery and deployment
  * Successful side branch catheterization and placement of bridging stents with restoration and maintenance of flow in all intended target vessels without the need for unanticipated corrective intervention related to placement of the bridging stent(s)
  * Successful withdrawal of the delivery systems without the need for unanticipated corrective intervention related to withdrawal
  * Absence of Type I or III endoleaks (assessed by Computed Tomography Angiography, Magnetic Resonance Angiography, or duplex ultrasound)
  * Patency of all aortic modular stent graft components

SECONDARY OUTCOMES:
All-Cause Mortality | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual component of the primary safety endpoint - defined as death due to any cause
Myocardial Infarction (new onset) | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual component of the primary safety endpoint - based on the SCAI definition
Respiratory failure | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual component of the primary safety endpoint - respiratory failure requiring prolonged (>24 hours from anticipated) mechanical ventilation or reintubation
Renal function decline | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual component of the primary safety endpoint - Renal function decline resulting in >50% reduction from baseline eGFR or new-onset dialysis
Bowel ischemia | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual component of the primary safety endpoint - Bowel ischemia requiring surgical resection or not resolving with medical therapy
Disabling stroke | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual component of the primary safety endpoint - Disabling stroke (mRS score ≥2 at 90 days post event and an increase in ≥1 mRS category from an individual's pre-stroke baseline, as direct result of the neurological event)
Paraplegia | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual component of the primary safety endpoint -Paraplegia grade 3, as per SVS TEVAR guidelines
Aneurysm-related mortality | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual components of the primary effectiveness endpoint - defined as death which occurs within the first 30-days of the index procedure or a secondary intervention, OR any death that results from aneurysm rupture or an aorta-related complication (e.g., implant infection, occlusion, dissection)
Aneurysm rupture | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual components of the primary effectiveness endpoint - Rupture of the native aneurysm sac (treated lesion)
Type I/III Endoleak | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual components of the primary effectiveness endpoint - Presence of Type I/IIIEndoleak as confirmed by imaging
Aneurysm Expansion | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual components of the primary effectiveness endpoint - Aneurysm expansion (>5 mm)
Device Migration | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual components of the primary effectiveness endpoint - Device migration (>10mm)
Loss of device patency | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual components of the primary effectiveness endpoint - complete occlusion of the aortic implant and/or bridging stent(s)
Conversion to open surgical repair | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual components of the primary effectiveness endpoint - Explant of the investigational device due to any cause
Secondary intervention (clinically significant) to address loss of patency, fixation or seal | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Individual components of the primary effectiveness endpoint. This includes the following reasons for re-intervention:
  Loss of Patency: Complete occlusion of the aortic endovascular graft, bridging stent(s), and/or limb(s) Seal: Type Ia/Ib, IIIa/IIIb/IIIc Endoleaks Fixation: Fracture, Kink, Migration Device System Prophylaxis: Device-related Reintervention requiring hospitalization
  Minor Secondary Interventions will not count against the endpoint and include the following:
  Endovascular procedures (completed for any reason), specifically percutaneous transluminal angioplasty, atherectomy, stenting without thrombectomy or thrombolysis Interventions to address branch vessel stenosis Interventions to address Type II endoleaks Minor surgical revisions (e.g., patch angioplasty) of the access vessel
Technical Success (at the index procedure) | At time of index procedure
  Technical Success (at the index procedure) is a composite of the following:
  * Successful access to the arterial system using remote arterial exposure, percutaneous technique, or open surgical conduit without the need for unanticipated corrective intervention related to access.
  * Successful delivery and deployment of the aortic stent-graft and all modular stent-graft components without the need for unanticipated corrective intervention related to delivery and deployment.
  * Successful side branch catheterization and placement of bridging stents with restoration and maintenance of flow in all intended target vessels without the need for unanticipated corrective intervention related to placement of the bridging stent(s)
  * Successful withdrawal of the delivery systems without the need for unanticipated corrective intervention related to withdrawal.
Presence of endoleak | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Evaluation of the presence of all endoleak types, as confirmed by imaging
Aneurysm size changes | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Evaluation of changes in aneurysm size. Enlargement is defined as >5mm, regression is ≥ 5 mm.
Device Migration Evaluation | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Evaluation of device migration. Migration is defined as >10mm.
Patency related observations | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Stenosis and occlusion of the components of the Fenestrated TREO Stent-Graft System
Loss of device integrity | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Fracture of stent strut, barb, or fenestration ring in Fenestrated TREO, fracture of stent in any Fenestrated TREO system implant
Target vessel instability | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Target vessel instability is a composite endpoint consisting of the following side branch complications:
  * Death related to side branch complication(s)
  * Rupture related to side branch complication(s)
  * Secondary intervention to address a side branch-related complication
Secondary interventions related to the device/treated lesion | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Any secondary interventions that are performed that are related to the device or the treated lesion will be recorded.
Target vessel complications | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Including dissection and/or perforation
Access-related complications | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  Access-related complications
Serious Adverse Events | Evaluated at all follow up visits which occur at the following timepoints: at discharge, 30 days post-procedure, six months post-procedure, 12-months post-procedure and annually thereafter through to five years post-procedure.
  As per protocol definition
Operative metrics - Time | Perioperative
  Information relating to the time of the surgical procedure such as start time, stop time, duration of procedure (min) and length of endovascular time (min)
Operative metrics - Number of Vessels intended to be Perfused via Fenestrated TREO Fenestrations | Evaluated at time of implant
  Information relating to the number and name of the vessels to be perfused via the Fenestrated TREO Fenestrations
Operative metrics - Mechanism of access | Evaluated at time of implant
  Information relating to the mechanism of access for the endovascular procedure
Radiation Exposure - Fluoroscopy Time | Evaluated at time of implant
  Fluoroscopy time (min)
Radiation Exposure - Total volume of Contrast | Evaluated at time of implant
  Volume of contrast used during procedure measured in mL

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Starnes, MD, Principal Investigator — University of Washington
Locations (5):
- United States (5):
  - Tampa General Hospital, Tampa, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Baylor Scott and White Research Institute, Plano, Texas
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Publications and presentations referring to the study will be coordinated by a Study Publication Committee overseen by the Sponsor. This committee will be responsible for the following activities: determining the scope of each publication; reviewing data provided by the Biostatistician; writing scientific papers or preparing presentation; submitting papers for publication or abstracts for conference/congress presentations. Decisions on IPD sharing will be taken as part of the study publication process.

REFERENCES:
- [Background] Starnes BW, Zettervall S, Larimore A, Singh N. Long-Term Results of Physician-Modified Endografts for the Treatment of Elective, Symptomatic, and Ruptured Juxtarenal Abdominal Aortic Aneurysms. Ann Surg. 2024 Oct 1;280(4):633-639. doi: 10.1097/SLA.0000000000006422. Epub 2024 Jun 26. PMID 38920026
- [Background] Tinelli G, Sica S, Sobocinski J, Ribreau Z, de Waure C, Ferraresi M, Snider F, Tshomba Y, Haulon S. Long-Term Propensity-Matched Comparison of Fenestrated Endovascular Aneurysm Repair and Open Surgical Repair of Complex Abdominal Aortic Aneurysms. J Endovasc Ther. 2024 Dec;31(6):1208-1217. doi: 10.1177/15266028231162256. Epub 2023 Mar 28. PMID 36978269
- [Background] Deery SE, Lancaster RT, Baril DT, Indes JE, Bertges DJ, Conrad MF, Cambria RP, Patel VI. Contemporary outcomes of open complex abdominal aortic aneurysm repair. J Vasc Surg. 2016 May;63(5):1195-200. doi: 10.1016/j.jvs.2015.12.038. PMID 27109792
- [Background] Locham S, Dakour-Aridi H, Bhela J, Nejim B, Bhavana Challa A, Malas M. Thirty-Day Outcomes of Fenestrated and Chimney Endovascular Repair and Open Repair of Juxtarenal, Pararenal, and Suprarenal Abdominal Aortic Aneurysms Using National Surgical Quality Initiative Program Database (2012-2016). Vasc Endovascular Surg. 2019 Apr;53(3):189-198. doi: 10.1177/1538574418819284. Epub 2018 Dec 26. PMID 30587096
- [Background] Meuli L, Kaufmann YL, Lattmann T, Attigah N, Dick F, Mujagic E, Papazoglou DD, Weiss S, Wyss TR, Zimmermann A. Editor's Choice - Peri-operative Mortality and Morbidity of Complex Abdominal Aortic Aneurysm Repair in Switzerland: A Swissvasc Report. Eur J Vasc Endovasc Surg. 2025 Jan;69(1):25-35. doi: 10.1016/j.ejvs.2024.06.022. Epub 2024 Jun 19. PMID 38906370
- [Background] Latz CA, Boitano L, Schwartz S, Swerdlow N, Dansey K, Varkevisser RRB, Patel V, Schermerhorn ML. Editor's Choice - Mortality is High Following Elective Open Repair of Complex Abdominal Aortic Aneurysms. Eur J Vasc Endovasc Surg. 2021 Jan;61(1):90-97. doi: 10.1016/j.ejvs.2020.09.002. Epub 2020 Oct 9. PMID 33046385
- [Background] Michel M, Becquemin JP, Clement MC, Marzelle J, Quelen C, Durand-Zaleski I; WINDOW Trial Participants. Editor's choice - thirty day outcomes and costs of fenestrated and branched stent grafts versus open repair for complex aortic aneurysms. Eur J Vasc Endovasc Surg. 2015 Aug;50(2):189-96. doi: 10.1016/j.ejvs.2015.04.012. Epub 2015 Jun 19. PMID 26100447
- [Background] Inker LA, Astor BC, Fox CH, Isakova T, Lash JP, Peralta CA, Kurella Tamura M, Feldman HI. KDOQI US commentary on the 2012 KDIGO clinical practice guideline for the evaluation and management of CKD. Am J Kidney Dis. 2014 May;63(5):713-35. doi: 10.1053/j.ajkd.2014.01.416. Epub 2014 Mar 16. PMID 24647050
- [Background] Vaidya SR, Aeddula NR. Chronic Renal Failure. In: StatPearls. Treasure Island (FL): StatPearls Publishing, http://www.ncbi.nlm.nih.gov/books/NBK535404/ (2023, accessed 18 September 2023)
- [Background] Moussa ID, Klein LW, Shah B, Mehran R, Mack MJ, Brilakis ES, Reilly JP, Zoghbi G, Holper E, Stone GW. Consideration of a new definition of clinically relevant myocardial infarction after coronary revascularization: an expert consensus document from the Society for Cardiovascular Angiography and Interventions (SCAI). J Am Coll Cardiol. 2013 Oct 22;62(17):1563-70. doi: 10.1016/j.jacc.2013.08.720. PMID 24135581
- [Background] Fillinger MF, Greenberg RK, McKinsey JF, Chaikof EL; Society for Vascular Surgery Ad Hoc Committee on TEVAR Reporting Standards. Reporting standards for thoracic endovascular aortic repair (TEVAR). J Vasc Surg. 2010 Oct;52(4):1022-33, 1033.e15. doi: 10.1016/j.jvs.2010.07.008. No abstract available. PMID 20888533
- [Background] Chaikof EL, Blankensteijn JD, Harris PL, White GH, Zarins CK, Bernhard VM, Matsumura JS, May J, Veith FJ, Fillinger MF, Rutherford RB, Kent KC; Ad Hoc Committee for Standardized Reporting Practices in Vascular Surgery of The Society for Vascular Surgery/American Association for Vascular Surgery. Reporting standards for endovascular aortic aneurysm repair. J Vasc Surg. 2002 May;35(5):1048-60. doi: 10.1067/mva.2002.123763. No abstract available. PMID 12021727
- [Background] Zettervall SL, Starnes BW. Planning and sizing of fenestrated/branched stent grafts. Semin Vasc Surg. 2022 Sep;35(3):252-258. doi: 10.1053/j.semvascsurg.2022.07.006. Epub 2022 Aug 6. PMID 36153066
- [Background] Lott A, Reiter JP. Wilson Confidence Intervals for Binomial Proportions With Multiple Imputation for Missing Data. The American Statistician 2020; 74: 109-115.
- [Background] Raulli SJ, Gomes VC, Parodi FE, Vasan P, Sun D, Marston WA, Pascarella L, McGinigle KL, Wood JC, Farber MA. Five-year outcomes of fenestrated and branched endovascular repair of complex aortic aneurysms based on aneurysm extent. J Vasc Surg. 2024 Aug;80(2):302-310. doi: 10.1016/j.jvs.2024.04.017. Epub 2024 Apr 10. PMID 38608964
- [Background] Hemingway JF, Starnes BW, Kline BR, Singh N. Initial experience with the Terumo aortic Treo device for fenestrated endovascular aneurysm repair. J Vasc Surg. 2021 Sep;74(3):823-831.e1. doi: 10.1016/j.jvs.2021.01.042. Epub 2021 Feb 14. PMID 33592291
- [Background] Nguyen T, Gittinger M, Gryzbowski C, Patel S, Asirwatham M, Grundy S, Zwiebel B, Shames M, Arnaoutakis DJ. One-hundred Consecutive Physician-Modified Fenestrated Endovascular Aneurysm Repair of Pararenal and Thoracoabdominal Aortic Aneurysms Using the Terumo TREO Stent Graft. Ann Vasc Surg. 2024 Sep;106:369-376. doi: 10.1016/j.avsg.2024.04.009. Epub 2024 May 31. PMID 38823478
- [Background] Yeung KK, Nederhoed JH, Tran BL, Di Gregorio S, Pratesi G, Bastianon M, Melani C, Riambau V, Bloemert-Tuin T, Hazenberg CEVB, van Herwaarden JA, Balm R, Lely RJ, van der Meijs BB, Blankensteijn JD, Hoksbergen AWJ, Jongkind V. Endovascular Repair of Juxtarenal and Pararenal Abdominal Aortic Aneurysms Using a Novel Low-Profile Fenestrated Custom-Made Endograft: Technical Details and Short-Term Outcomes. J Endovasc Ther. 2025 Dec;32(6):1988-1993. doi: 10.1177/15266028241227392. Epub 2024 Jan 30. PMID 38288587
- [Background] Eagleton MJ, Stoner M, Henretta J, Dryjski M, Panneton J, Tassiopoulos A, Mehta M, Pearce B, Sharafuddin MJ; TREO Investigators. Safety and effectiveness of the TREO stent graft for the endovascular treatment of abdominal aortic aneurysms. J Vasc Surg. 2021 Jul;74(1):114-123.e3. doi: 10.1016/j.jvs.2020.10.083. Epub 2020 Nov 28. PMID 33253871
- [Background] Oderich GS, Forbes TL, Chaer R, Davies MG, Lindsay TF, Mastracci T, Singh MJ, Timaran C, Woo EY; Writing Committee Group. Reporting standards for endovascular aortic repair of aneurysms involving the renal-mesenteric arteries. J Vasc Surg. 2021 Jan;73(1S):4S-52S. doi: 10.1016/j.jvs.2020.06.011. Epub 2020 Jun 29. PMID 32615285